CLINICAL TRIAL: NCT01482468
Title: Effect of Continuous Infusion of Palonosetron Following Single Prophylactic Injection of Palonosetron for Preventing Postoperative Nausea and Vomiting
Brief Title: Continuous Infusion of Palonosetron for Preventing of Postoperative Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Soo Kyoung Park, Clnical professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OC11MISI0109
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous infusion (Active Comparator): continuous infusion of palonosetron added to prophylactic single injection of palonosetron
  Interventions: Drug: continuous infusion of palonosetron added to prophylactic single injection of palonosetron
- singel injection (Placebo Comparator): continuous infusion of normal saline added to prophylactic single injection of palonosetron
  Interventions: Drug: continuous infusion of normal saline added to prophylactic single injection of palonosetron

INTERVENTIONS:
Drug: continuous infusion of palonosetron added to prophylactic single injection of palonosetron — continuous infusion of palonosetron 0.00075 mg/hour after single injection of palonosetron 0.075mg
  Arms: continuous infusion
Drug: continuous infusion of normal saline added to prophylactic single injection of palonosetron — continuous infusion of normal saline after single injection of palonosetron 0.075mg
  Arms: singel injection

SUMMARY:
The purpose of this study is to determine whether continuous infusion of palonosetron after its prophylactic single injection can further reduce the incidence of postoperative nausea and vomiting in patients undergoing gynecological laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1 or 2
* Elective gynaecological laparoscopic surgery of ≥ 1h duration

Exclusion Criteria:

* Anti-emetics, steroids, or psychoactive medications within 24 h of study initiation
* Vomiting or retching in the 24 h preceding surgery
* Cancer chemotherapy within 4 weeks or emetogenic radiotherapy within 8 weeks before study entry
* Ongoing vomiting from gastrointestinal disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | 24 hours after surgery

SECONDARY OUTCOMES:
severity of nausea | for 24 hours after sugery

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St Mary's hospital, Incheon, South Korea